CLINICAL TRIAL: NCT04978272
Title: Enhancing Immunity to Malaria in Young Children With Effective Chemoprevention
Brief Title: Modifying Immunity in Children With DihydROartemisinin-Piperaquine (MIC-DroP)
Acronym: MIC-DroP
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Grant Dorsey, M.D, Ph.D. (Other)
Collaborators: Stanford University (Other); Infectious Diseases Research Collaboration, Uganda (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Karolinska Institutet (Other)
Responsible Party: Sponsor-Investigator, Grant Dorsey, M.D, Ph.D., Professor, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Prevention
Other Study IDs: MIC-DroP; U01AI155325 (NIH)
Record Dates: First submitted 2021-07-23; First posted 2021-07-27 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Malaria
Keywords: dihydroartemisinin-piperaquine; intermittent preventive therapy; children; immune response
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Intervention Model Description: Double blinded randomized controlled trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: Administration of all study drugs will be double blinded. All doses of study drugs will be prepackaged by a study pharmacist and administered by a study nurse blinded to the study participant's treatment regimen. All 3 daily doses will be directly observed in the clinic. If a study participant vomits the study drug within 30 minutes of administration, the drug will be re-administered. All doses of study drugs will be given between 8 and 104 weeks (2 years) of age.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- IPTc DP 1 year (Active Comparator): DP given from 8 weeks to 52 weeks of age; DP placebo given from 52 weeks to 104 weeks of age; No IPTc in third and fourth years of follow-up.
  Interventions: Drug: Dihydroartemisinin-piperaquine (DP); Other: DP Placebo
- IPTc DP 2 years (Active Comparator): DP given from 8 weeks to 104 weeks of age; No IPTc in third and fourth years of follow-up.
  Interventions: Drug: Dihydroartemisinin-piperaquine (DP)
- No IPTc (Placebo Comparator): DP placebo given from 8 weeks to 104 weeks of age; No IPTc in third and fourth years of follow-up.
  Interventions: Other: DP Placebo

INTERVENTIONS:
Drug: Dihydroartemisinin-piperaquine (DP) — Duo-Cotecxin 20mg/160mg tabs by Holley-Cotec, Beijing, China Each treatment with DP will consist of half-strength tablets given once a day for 3 consecutive days according to weight-based guidelines.
  Other Names: Duo-Cotecxin
  Arms: IPTc DP 1 year; IPTc DP 2 years
Other: DP Placebo — Placebos will be identical appearance to DP.
  Arms: IPTc DP 1 year; No IPTc

SUMMARY:
The MIC-DroP trial will test the hypothesis that preventing early life blood-stage malaria antigenic exposure with intermittent preventive therapy (IPT) enhances protective immunity to malaria. This study will take advantage of a unique opportunity to study infants born to mothers followed in a NIH-funded randomized controlled trial of novel intermittent preventive therapy in pregnancy (IPTp) regimens (NCT04336189). MIC-DroP will leverage the parent IPTp study to enroll 924 children who will be randomized at 8 weeks of age to receive no intermittent preventive therapy in childhood (IPTc), monthly DP from 8 weeks to 1 year of age, or monthly DP from 8 weeks to 2 years of age, and then follow children to 4 years of age. The primary outcome of this study will be to compare the incidence of malaria from 2 to 4 years of age among children randomized to receive no IPTc, monthly DP for the first year of life, or monthly DP for the first two years of life. Investigators will also leverage this trial to evaluate immune development during early childhood.

DETAILED DESCRIPTION:
This study is a phase III, double-blind, randomized controlled trial of 924 HIV- uninfected children. Children born to mothers enrolled in an ongoing clinical trial of different IPTp arms in pregnancy (NCT 04336189) will be enrolled in this study. In the parent IPTp study, 2757 HIV-uninfected pregnant women will be randomized to receive IPTp with monthly sulfadoxine pyrimethamine (SP) alone, monthly DP alone, or both monthly SP+DP, and followed through 4 weeks postpartum. At the 4-week postpartum visit, we will enroll and randomize 924 eligible children to one of three IPTc arms: no IPTc (the current standard of care), monthly DP from 8 weeks to 1 year of age, or monthly DP from 8 weeks to 2 years of age. Study drugs will be placebo controlled and all doses of study drug will be given by directly observed therapy (DOT). The intervention phase will be completed at 2 years of age, and children followed through 4 years of age. Study participants will be followed for all of their outpatient medical care in our dedicated study clinic. Malaria incidence will be measured via active case detection. Routine assessments will be performed in the study clinic for all study participants every 4 weeks, including passive surveillance for parasitemia by quantitive polymerase chain reaction (qPCR). Venous blood will be collected for immunologic assays three times annually from 8 weeks to 4 years of age. All maternal assessments conducted during the parent IPTp study, including assessment for maternal malaria exposure (e.g., placental histology) household survey, will be available and linked to each study participant.

ELIGIBILITY:
Inclusion Criteria:

1. Born to HIV-uninfected mother enrolled in parent clinical trial of intermittent preventative treatment of malaria in pregnancy (IPTp-SP vs. IPTp-DP vs. IPTp-SP+DP, NCT 04336189)
2. Resident of Busia District
3. Provision of informed consent by parent/guardian
4. Agreement to present for any illness and avoid, where possible, medications outside the study protocol.

Exclusion Criteria:

1. Intention of moving outside Busia district during the study period
2. Active medical problem requiring in-patient evaluation or chronic medical condition requiring frequent medical attention

Max Age: 2 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 924 (Actual)
Dates: Start 2022-02-08 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of symptomatic malaria following cessation of IPTc | 2 years to 4 years of age
  The incidence of symptomatic malaria, defined as the number of incident episodes of malaria requiring treatment per time at risk, during the period after the intervention was given (2-4 years of age). Treatments within 14 days of a prior episode are not considered incident events.

SECONDARY OUTCOMES:
Incidence of complicated malaria | 2 years to 4 years of age
  Any incident episode of malaria meeting World Health Organization criteria for severe malaria or danger signs per time at risk, during the period after the intervention was given (2-4 years of age).
Incidence of hospital admissions and/or deaths | 2 years to 4 years of age
  Admission to the pediatric ward for any cause, and deaths of any cause
Prevalence of parasitemia | 2 years to 4 years of age
  Proportion of routine visits with asexual parasites detected by blood smears or quantitative polymerase chain reaction (qPCR).
Prevalence of anemia | 2 years to 4 years of age
  Proportion of routine hemoglobin measurements <11 grams/dL

CONTACTS AND LOCATIONS:
Overall Officials: Prasanna Jagannathan, MD, Principal Investigator — Stanford University
Locations (1):
- IDRC - Tororo Research Clinic, Tororo, Uganda

IPD SHARING:
Plan to Share IPD: No